CLINICAL TRIAL: NCT06085911
Title: Intervention Against Long COVID in Norway - Systematic Rehabilitation. A Randomised Pilot and Feasibility Study.
Brief Title: RCT Long COVID-19 Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Bergen (Other); Oslo University Hospital (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 587293
Record Dates: First submitted 2023-10-16; First posted 2023-10-17 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2023-09

CONDITIONS: Rehabilitation; Post-Acute COVID-19 Syndrome; Post-Infectious Disorders
Keywords: Rehabilitation; Long COVID; Clinical trial; Telemedicine; Inflammation; Post-Acute COVID-19 Syndrome; COVID-19; Post-Infectious Disorders
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Post-Infectious Disorders; Inflammation; COVID-19

STUDY DESIGN:
Intervention Model Description: randomized controlled trial (RCT) comparing two intervention groups
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- individual follow-ups (Experimental): tailored individual follow-up rehabilitation program with home-based exercises
  Interventions: Behavioral: Individual follow-ups
- a one-day course. (Active Comparator): a one-day course.
  Interventions: Behavioral: One day course

INTERVENTIONS:
Behavioral: One day course — a physical one-day course at the Covid rehabilitation clinic. During these six hours, general information about rehabilitation principals will be given. Theory about three 15 focus areas of importance will be presented; daily routine, importance of being active and cognitive training. They will meet others with similar problems and will be given an opportunity to exchange experience. 8-10 patients will participate in the group.
  Arms: a one-day course.
Behavioral: Individual follow-ups — the patient will meet a therapist in a physical consultation at the Covid rehabilitation clinic lasting for 1.5 hours. Together they will in detail map out symptoms and impairment of function in the patient's life. Together the patient and the therapist will create plan to address these problems consisting of tailored home-based exercises within the three focus areas. Tree follow-up consultations will be given.
  Arms: individual follow-ups

SUMMARY:
The Coronavirus 2019 (COVID-19) pandemic has resulted in at least four million infections in Norway. The vast majority of cases are diagnosed and followed up in the community, but some with extensive symptoms and large degree of reduced function are referred to regional Covid-clinics. In total this patient group is placing an enormous burden on the already over stretched health care services. As the pandemic subsides the emerging threat of long-term disability from COVID remains to be quantified. Brain fog and cognitive symptoms are common in long COVID in 30% of mild infections resulting in sick leave and loss of daily function, with women overrepresented among long COVID sufferers. The true prevalence and underlying mechanisms of long COVID remains to be quantified. Although vaccination prevents severe infection and death, we have little knowledge on how best to rehabilitate those who suffers from long COVID.

Here we propose to develop knowledge on treatment interventions to counteract disability from long COVID and lessening the burden on health care services. We will conduct a study of where we compare a short group intervention with systematic personalised neurocognitive rehabilitation to document symptom alleviation. Our overarching goal is to develop effective programmes for this evolving disease to reduce the suffering for the patients, and thereby reducing costs for health services and society at large.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms attributable to long COVID according to WHO definition [14] that affect their daily activities
* Positive Covid test; a home-test, PCR test or serology.
* Neurocognitive symptoms
* Age between 18 and 65 years
* Participant is able and willing to provide informed consent

Exclusion Criteria:

* Patients that do not want to comply to planned physical study visits
* Patients who are unable to complete surveys in Norwegian
* Patients with known chronic neurocognitive disease before Covid-19 or other diseases that can explain current symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Symptom reduction | 3 months
  A reduction in number present symptoms is evaluated in each patient group. A significant greater alleviation in the of number symptoms at three months is considered as a better prognosis.

SECONDARY OUTCOMES:
Symptoms grouped by systems reduction | 12 month follow-up
  All individual symptoms separately, and grouped by systems (systemic symptoms, chest-symptoms, cognitive, other neurocognitive symptoms) and as full recovery (absence of all symptoms) at 3-, 6- and 12 months.
Graded symptom reduction | 3-12 months
  Graded responses for separate symptoms and symptom constellations, including an ordinal variable graded 0-3 for the presence of neurocognitive relevant symptoms and dyspnea.
Work improvement | 3-12 months
  Improvement in work participation
Quality of life improvement | 3-12 months
  Improvement in quality of life measured by EQ-5D-5L and measurement of Quality-adjusted life year (QALY)
Neuropsychological functions improvement | 6 months
  Improvement of neuropsychological functions

CONTACTS AND LOCATIONS:
Overall Officials: Maja Wilhelmsen, ph.d, Principal Investigator — University Hospital of North Norway
Locations (1):
- University hospital of North Norway, Tromsø, Troms, Norway